CLINICAL TRIAL: NCT00761553
Title: Dietary Supplements and Exercise in Aging Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Wayne Campbell, Ph.D., Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0509003026; NIH/NIA 5R01AG021911
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Exercise
Keywords: The study is designed to determine the effects of food supplements and strength training.
MeSH Terms: conditions — Motor Activity | interventions — Dietary Supplements; Exercise

ARMS (4):
- 1 (Experimental): Solid dietary supplements with exercise
  Interventions: Other: Dietary supplements with exercise
- 2 (Experimental): Solid dietary supplements without exercise
  Interventions: Dietary Supplement: Dietary supplement without exercise
- 3 (Experimental): Liquid dietary supplements with exercise
  Interventions: Other: Dietary supplements with exercise
- 4 (Experimental): Liquid supplements without exercise
  Interventions: Dietary Supplement: Dietary supplement without exercise

INTERVENTIONS:
Other: Dietary supplements with exercise — Resistive exercise along with consuming two dietary supplements every day during both 8 week intervention periods, for a total of 16 weeks.
  Arms: 1; 3
Dietary Supplement: Dietary supplement without exercise — Consuming two dietary supplements every day during both 8 week intervention periods, for a total of 16 weeks.
  Arms: 2; 4

SUMMARY:
The purpose of this study is to determine the effects of food supplements and strength training on appetite, the amount of energy used, and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 55 and older
* Body mass index 20 to ≤35 kg/m2
* Weight stable (<4kg change within the last 3 months)
* Constant habitual activity patterns (no deviation > 1x/wk of 30 min/session within last 3 months)
* Clinically normal blood and urine profiles as determined by our study physician
* Not taking medications known to influence appetite nor any anti-inflammatory steroid medications
* No hip replacements

Exclusion Criteria:

* Adults with medical conditions that might place them at risk for participating in the study or interfere with the successful completion of the study protocol will be excluded

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Appetite questionnaire, urine collection, strength testing, body composition, resting metabolic rate, food records, breath sample, activity assessments, dietary supplements, nightly logs, and resistive exercise. | 23 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States